CLINICAL TRIAL: NCT00329511
Title: A Comparison of Compliance Between Clonidine Patch and Methyldopa for the Treatment of Chronic Hypertension in Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility of study. PI termination
Sponsor: Afshan B. Hameed, M.D. (Other)
Responsible Party: Sponsor-Investigator, Afshan B. Hameed, M.D., Associate Professor, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200-04
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: pregnancy; hypertension; compliance; clonidine patch; methyldopa
MeSH Terms: conditions — Hypertension; Patient Compliance | interventions — Methyldopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): methyldopa
  Interventions: Drug: methyldopa vs. clonidine; Drug: clonidine patch
- B (Active Comparator): clonidine patch
  Interventions: Drug: methyldopa vs. clonidine; Drug: clonidine patch

INTERVENTIONS:
Drug: methyldopa vs. clonidine — Comparison of compliance
Drug: clonidine patch — methyldopa 250 - 750 mg qid clonidine patch 0.1 - 0.4 mg q week
  Other Names: aldomet; catapress tts

SUMMARY:
High blood pressure (BP) before pregnancy is called chronic hypertension (CHTN), and is associated with an increased risk of development of pregnancy related high BP called preeclampsia, preterm delivery, decreased growth of the fetus, fetal death, premature separation of the placenta from the uterus resulting in damage to the fetus and cesarean delivery. Longer duration and severity of CHTN in pregnancy leads to worse outcomes for the mother and the fetus. Treatment of mild CHTN in pregnancy does not improve these outcomes, and therefore, medications to lower BP are used for moderate to severe hypertension. To date the literature on the medications used in pregnancy is extremely limited.

Methyldopa is used as a first choice medicine for CHTN in pregnancy. It acts on the central nervous system (CNS) by relaxation of the blood vessels leading to a decrease in BP. It does not decrease the blood flow to the uterus, placenta, or the fetus (4). Methyldopa is a weak antihypertensive medicine given three or four times a day and frequently needs changes in the dose or may require an additional medication to control BP. This may lead to a greater chance of non compliance. Another option is Clonidine which is an effective antihypertensive treatment and is available in many forms (oral, parenteral, and transdermal.) It acts on the maternal CNS. Clonidine is not associated with teratogenic or neonatal side effects. Transdermal clonidine (catapres-TTS®) is a preparation of clonidine hydrochloride that can be released and absorbed transdermally over a 7-day period.

The study will determine differences in compliance between the two antihypertensive regimens- oral methyldopa and Catapres-TTS, comparisons of patient tolerability, compliance and adequacy of BP control, as well as provide information on an alternate option for BP control.

DETAILED DESCRIPTION:
Purpose of the Study:

The purpose of this of open-label randomized clinical trial is to compare clonidine patch (Catapres-TTS®) and orally administered methyldopa (Aldomet®) over a 4-week period for compliance in pregnant women between 14 and 28 weeks of gestation. In addition, this study will evaluate blood pressure (BP) control, patient tolerability, and development of side effects to each medication. Patients will be alternately randomized to receive methyldopa (standard of care) or clonidine patch.

Hypothesis:

Clonidine is an effective antihypertensive agent with similar mechanism of action to methyldopa. Transdermal clonidine may provide a better compliance profile, adequate BP control and, therefore, may be used as an alternative to methyldopa for the treatment of CHTN in pregnancy.

Primary outcome of the study is patient compliance. Compliance will be measured via patient diary, promptness of keeping appointments, and pill/patch counts at each visit. Overall compliance will be calculated over a 4 week study period by adding compliance points for each visit as outlined in the data sheet.

Secondary outcomes are:

1. Change in mean arterial BP at weeks 1,2,3,4 in comparison to baseline BP at the initial visit (It will be used in patients newly started on medications or in patients with uncontrolled BP at baseline).
2. Side effects to each medication as reported by the patients.

Background and Significance

Chronic hypertension (CHTN) affects 1-5% of pregnancies. It is defined as BP of 140/90 or higher before the 20th week of gestation or beyond 12 weeks postpartum. CHTN is associated with an increased risk of preeclampsia, preterm delivery, intrauterine growth restriction, intrauterine fetal demise, placental abruption and cesarean delivery. Mild hypertension is defined as BP < 150/100 mm Hg and severe hypertension as BP > 160/110 mm Hg. There is a direct correlation of adverse perinatal outcomes with duration and severity of CHTN in pregnancy. Treatment of mild CHTN in pregnancy does not improve perinatal outcomes, and therefore, antihypertensive therapy is reserved for moderate to severe hypertension only.

Methyldopa is used as a first line therapy for CHTN in pregnancy. It is a central alpha-adrenergic agonist that decreases peripheral sympathetic outflow and thus results in a decrease in peripheral resistance and BP. It does not impact uteroplacental blood flow and fetal hemodynamics. Methyldopa is a weak antihypertensive agent and often times there is a need for increase in dose, frequency and/or addition of another medication to optimize BP control with advancing gestational age. Side effects of methyldopa include sedation, orthostatic hypotension, edema, weight gain, bradycardia, and dry mouth. Rarely, aggravation of angina, congestive heart failure, pancreatitis, colitis, hyperprolactinemia, bone marrow depression, hemolytic anemia, false positive anti-nuclear antibodies and rheumatoid factor may be seen.

The use of various classes of antihypertensive medications in pregnancy is limited due to potential teratogenic effects. Angiotensin converting enzyme inhibitors are contraindicated in pregnancy. The use of beta-blockers and diuretics is controversial, and there is limited data on calcium channel blockers in pregnancy.

Clonidine is an effective antihypertensive treatment and is available in oral, parenteral, and transdermal dosage forms. Although oral and parenteral forms are commonly employed for short-term use in hypertensive urgencies, data regarding its use in pregnancy are lacking. It acts by stimulating α2-adrenergic receptors in the central nervous system (CNS), which depresses peripheral sympathetic nervous system outflow, and thus lowering BP. Clonidine is not associated with teratogenic effects in the fetus. Reproduction studies performed in rabbits at doses up to 3 times the maximum recommended daily human dose (MRDHD) of clonidine hydrochloride have revealed no evidence of teratogenic or embryotoxic potential. The pharmacokinetics of clonidine in pregnancy has been studied. Clonidine crossed placenta and fetal concentration is 0.89 of the maternal level. No neonatal side effects have been reported. Clonidine is metabolized by the liver and is excreted unchanged in the urine.

Therapeutic levels of orally administered drugs are affected by the transit time through small intestines and the presence of food and liquid in the gastrointestinal tract. Transdermal administration of drugs by passes the first-pass metabolism through the liver, requires smaller dose to achieve therapeutic effects, and promotes patient compliance. In addition, the drug is absorbed through the skin at a constant rate eliminating peak and troughs associated with oral administration. This may result in steadier BP control with transdermal clonidine administration. This may be of benefit in pregnancy as the gastrointestinal transit time is significantly prolonged due to progesterone effects and nausea vomiting in the first trimester may limit the use of orally administered drugs. In addition, one would expect improved patient compliance be avoiding repeated dosing such as four times a day schedule for methyldopa.

Transdermal clonidine (Catapres-TTS®) is a preparation of clonidine hydrochloride that can be released and absorbed transdermally over a 7-day period. Its side effect profile is similar to methyldopa including tiredness, lethargy, drowsiness, constipation and dry mouth. Orthostatic hypotension occurs in 3% patients with oral administration and has not been reported with the transdermal form. Skin reactions including redness, itching, and darkening of the skin may occur with clonidine patches. Rarely, angioedema, atrioventricular block, chest pain, congestive heart failure, hepatitis, thrombocytopenia, or urinary retention may occur.

A study of hypertension in non-pregnant individuals from United Kingdom showed that only 40% of patients who were started on a new antihypertensive drug were compliant six months later. There are no data available on compliance with antihypertensive medications in pregnancy, although our anecdotal experience is of improved compliance with medications in pregnancy compared to a non-pregnant state.

Our study will determine differences in compliance between the two antihypertensive drugs, and will provide additional comparisons of patient tolerability and adequacy of BP control. This may be of particular value in pregnant women who are unable to tolerate oral feeds e.g. those with hyperemesis gravidarum, or in immediate postoperative period. In addition, it will provide information on an alternate option for BP control, which has not been described in obstetrical literature.

1. National High Blood Pressure Educational Program Working Group. Report on High Blood Pressure in Pregnancy. Am J Obstet Gynecol 1990;163:1691-1712.
2. Report of the National High Blood Pressure Education Program Working Group on High Blood Pressure in Pregnancy. Am J Obstet Gynecol 2000;183:S1-S22.
3. Chronic Hypertension in Pregnancy. ACOG Practice Bulletin No. 29. American College of Obstetricians and Gynecologists. Obstet Gynecol 2001;98:177-185.
4. Montan S, Anandakumar C, Arulkumaran S, Ingemarsson I, Ratnam SS. Effects of Methyldopa on Uteroplacental and Fetal Hemodynamics in Pregnancy Induced Hypertension. Am J Obstet Gynecol 1993;168:152-6.
5. Horrath JS, Phippard A, Korda A, Hendersen-Sart DJ, Child A, Tiller DJ. Clonidine Hydrochloride - A Safe and Effective Antihypertensive in Pregnancy. Obstet Gynecol 1985;66:634-8.
6. Turnbull AC, Ahmad S. Catapress in the Treatment of Hypertension in Pregnancy, A Preliminary Study. In Hypertension. Symposium of the Royal College of Surgeons, London 1970:237-45
7. Hartikainen-Sorri AL, Heikkinen JE, Koivisto M. Pharmacokinetics of Clonidine During Pregnancy and Nursing. Obstet Gynecol 1987;69:598-600.
8. Ala-Kokko TI, Pienimaki P, Lampela E, Hollmen AI, Pelkonen O, Vahakangas K. Transfer of Clonidine and Dexmedetrmidine Across the Isolated Perfused Human Placenta. Acta Anesthesiol Scand 1997;41(2):313-19.
9. Jones JK, Gorkin L, Lian JF, Staffa JA, Fletcher AP. Discontinuation of and Changes in Treatment after start of new courses of Antihypertensive Drugs: A Study of a United Kingdom Population. BMJ 1995;311:293-5

ELIGIBILITY:
Inclusion Criteria:

1. Intrauterine pregnancy between 14 - 28 weeks of gestation
2. Chronic hypertension requiring antihypertensive therapy (BP < 180/110)
3. Subjects who consent to the study
4. No evidence of fetal compromise (i.e. intrauterine growth restriction)

Exclusion Criteria:

1. Evidence or suspicion of preeclampsia
2. Known cardiac disease
3. Known renal dysfunction (creatinine > 1 mg/dl)
4. Known hepatic disease
5. Known cerebrovascular disease
6. Allergy to clonidine patch

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Comparison of compliance | 4 weeks

SECONDARY OUTCOMES:
Side effects | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Afshan B Hameed, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States